CLINICAL TRIAL: NCT03144726
Title: Single Center Prospective Randomized Control Trial on Negative Pressure Wound Therapy for Incisions Following Major Lower-limb Amputation to Reduce Surgical Site Infection
Brief Title: RCT on NPWT for Incisions Following Major Lower-limb Amputation to Reduce Surgical Site Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Adam Power, Physician, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB 109128
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Amputation Wound; Amputation Stump Complication; Amputation Stump; Infection; Infection
MeSH Terms: conditions — Infections | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative pressure wound therapy (Experimental): A vacuum assisted closure device will be applied in this arm
  Interventions: Device: Negative pressure wound therapy
- Standard dressing (Other): Standard dressing will be applied to this arm
  Interventions: Other: Standard dressing

INTERVENTIONS:
Device: Negative pressure wound therapy — Negative pressure wound therapy is a commonly utilized tool in the hospital setting and will be applied to amputations in our study to determine the effect on surgical site infections
  Arms: Negative pressure wound therapy
Other: Standard dressing — A standard dressing will be applied to the amputations in this arm of the study
  Arms: Standard dressing

SUMMARY:
Surgical site infections following lower extremity amputations have been reported in up to 40% of patients. Surgical site infections have significant morbidity and even mortality in terms of emergency room visits, length of hospital stay, reamputation rates and death. Since its introduction, negative pressure wound therapy has been demonstrated to promote wound healing and possibly decreasing the need for future amputations. The aim of the study is to provide level I evidence for the use of negative pressure wound therapy devices in patients undergoing lower extremity amputation.

DETAILED DESCRIPTION:
Amputations are common vascular surgery procedures performed on patients with multiple medical comorbidities. Historically, morbidity and mortality following major amputation of the lower extremity in this patient population has been high. Recent studies have cited 30-day mortality rates ranging from 6% to 17%, with greater risk among patients with transfemoral vs transtibial amputation. Postoperative goals after amputation include uncomplicated wound healing and, for appropriate candidates, progression to use of a prosthesis for ambulation or transfer. Perioperative wound complications can be devastating in this already debilitated population and can range from 13% to 40%.

Postoperative wound complications, such as infection, dehiscence, and formation of haematoma or seroma, are common complications of surgical procedures; particularly among patients with risk factors such as obesity and diabetes. Wound complications may delay recovery, increase patient discomfort and reduce overall quality of life. Increased healthcare costs may be incurred due to prolonged inpatient stay, repeat surgery and the need for increased follow-up.

Wounds that are secondary to amputation are reported in 13-40% of cases and are one of the most challenging types of lower extremity wounds to heal. These patients often have compromised healing capacity. Kayssi et al studied Canadian readmission rates, early (<30 days) and late (30-365) readmissions were attributed to stump complications in 13% and 10% of patients respectively.

Wound complications in major limb amputation frequently result in the need for further major surgery in a group of patients with significant co-morbidity and enhanced operative risk. 1, 3, and 5 year reamputation rates for diabetics who have had major amputations are 4.7%, 11.8%, and 13.3% respectively. Henry et al suggested that undergoing multiple amputation revisions may indicate aggressive measures to treat critical limb ischemia or chronic infection that precede conversion to a more proximal amputation. Kono et al studied the incidence and risk factors for reamputation after forefoot amputation. They found that 16/116 (14%) patients developed postoperative infection, and 10 of these required reamputation (62.5%). Five of the ten reamputations occurred within 30 days after the patients developed postoperative infections.

In addition to the morbidity from infection there is also an increased rate of phantom pain as well as a delay to mobilisation with prosthesis. Minimizing postoperative infections would likely have improvements in clinical outcomes, quality of life, and utilization of resources. Currently, all patients are given prophylactic broad spectrum antibiotics to reduce the incidence of wound infection. Sadat et al investigated whether a prolonged 5 day course of antibiotics wound reduce stump infections, their results were positive however this treatment is associated with the increased risk of antimicrobial resistance and c. difficile infection.

Negative-pressure wound therapy (NPWT) has traditionally been used for the treatment of open wounds. In recent years, the indication for NPWT has been extended to include treatment of closed surgical incisions. Armstrong et al conducted a randomized controlled trial to determine whether NPWT delivered by the VAC system was clinically efficacious in treating amputation wounds of the diabetic foot to improve the proportion of wounds with complete closure. Treatment with NPWT resulted in a higher proportion of wounds that healed, faster healing rates, and fewer re-amputations than with standard treatment. No randomized controlled trials have been performed to assess NPWT and infection rates after major lower limb amputation.

There is a paucity of scientific literature reporting outcomes following major amputation in patients with critical limb ischemia, particularly with regards to wound problems and infection. The purpose of this study is to provide Level I evidence on whether negative pressure wound therapy is an effective strategy to significantly reduce postoperative infections after major lower extremity amputation, thereby reducing patient morbidity and mortality from this procedure.

ELIGIBILITY:
Inclusion Criteria:

* any patient 18 years or older undergoing amputation of the lower limb, either an above knee amputation (AKA) or below knee amputation (BKA)
* ability to read and write English to undergo informed consent

Exclusion Criteria:

* patients in which a complete seal cannot be obtained at the time of vacuum placement
* wounds that are not closed primarily
* existing infection
* patient is anticipated to not follow-up
* inability to read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Surgical site infection will be defined using the Centre for Disease Control and Prevention Guidelines.

SECONDARY OUTCOMES:
Length of stay | 30 days
  length of hospital stay
Antibiotic use | 30 days
  requirement for antibiotics to treat surgical site infection
Reoperation | 30 days
  requirement for revision of amputation
Death | 30 days
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Adam Power, MD, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: Undecided